CLINICAL TRIAL: NCT01331486
Title: Nitric Oxide Mediated Vasodilatory Response to Hawthorn Standardized Extract
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 09-2279
Record Dates: First submitted 2011-04-06; First posted 2011-04-08 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2011-12

CONDITIONS: Prehypertension; Mild Hypertension
Keywords: Prehypertension; Mild hypertension; Flow mediated dilation; Hawthorn
MeSH Terms: conditions — Prehypertension | interventions — crataegus extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo capsule
- Low dose (Active Comparator)
  Interventions: Dietary Supplement: Hawthorn
- Mid dose (Active Comparator)
  Interventions: Dietary Supplement: Hawthorn
- High dose (Active Comparator)
  Interventions: Dietary Supplement: Hawthorn

INTERVENTIONS:
Dietary Supplement: Hawthorn — Hawthorn standardized extract liquid capsule
  Other Names: Gaia Hawthorn Supreme
  Arms: High dose; Low dose; Mid dose
Dietary Supplement: Placebo capsule — Matched placebo liquid capsule
  Arms: Placebo

SUMMARY:
Prehypertension and mild hypertension affect an estimated 157 million U.S. adults. Cardiovascular disease (CVD) risk and associated mortality is elevated in this population. Treatment options are limited consisting of lifestyle modification, which is often ineffective, or drug therapy, which carries risk of side effects. Highly safe, efficacious, and acceptable treatment options for this population are needed. Hawthorn standardized extract (HSE) is approved for use in Europe to treat heart failure, and preliminary evidence suggests it may have a blood pressure lowering effect. However, prior trials of hawthorn have based dosage recommendations on animal studies. Therefore, the investigators propose a dose-finding study to measure the pharmacodynamic effect of three doses of standardized hawthorn extract and placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Recent ambulatory daytime systolic BP average between 120 - 155 mmHg or diastolic BP between 80-95 mmHg
2. Age 18 years and older.
3. Ability to speak English

Exclusion Criteria:

1. Any antihypertensive medication use (ACE inhibitors, ARB, beta-blockers, calcium channel blockers, diuretics, alpha agonists or antagonists, nitrates, direct vasodilators such as hydralazine, aldosterone antagonists, direct renin inhibitors, endothelin antagonists)
2. Current tobacco use.
3. Diagnosed with diabetes, known coronary artery disease, severe aortic stenosis, idiopathic hypertrophic subaortic stenosis (IHSS), or upper extremity vascular obstruction.
4. Pregnancy or breast feeding.
5. Using estrogen-containing birth control methods.
6. Unwillingness to forgo vitamins C and E, fish oil, niacin, arginine, OTC decongestants, and NSAIDs such as advil, motrin, and nuprin during the study period.
7. Unwillingness to forgo use of phosphodiesterase inhibitors (sildenafil - 36 hours, vardenafil - 36 hours, tadalafil - 96 hours) prior to study visits.
8. Unwillingness to refrain from vigorous exercise on the morning of study visits.
9. Women with childbearing potential who do not agree to practice effective birth control (condom, diaphragm, cervical cap, copper IUD, abstinence).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
FMD Max | 7d
  Brachial artery flow mediated dilation max (%)

SECONDARY OUTCOMES:
BP | 7d
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Gary N Asher, MD, MPH, Principal Investigator — UNC
Locations (1):
- UNC Department of Family Medicine, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Asher GN, Viera AJ, Weaver MA, Dominik R, Caughey M, Hinderliter AL. Effect of hawthorn standardized extract on flow mediated dilation in prehypertensive and mildly hypertensive adults: a randomized, controlled cross-over trial. BMC Complement Altern Med. 2012 Mar 29;12:26. doi: 10.1186/1472-6882-12-26. PMID 22458601